CLINICAL TRIAL: NCT03566784
Title: Electrocoagulation Employment During TAPP (Transabdominal Preperitoneal Approach) Inguinal Hernia Repair
Brief Title: Electrocoagulation Employment During TAPP Inguinal Hernia Repair
Status: Completed | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Other Study IDs: CHIR-02-Electrocoagulation
Record Dates: First submitted 2018-06-12; First posted 2018-06-25 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Inguinal Hernia
Keywords: inguinal hernia repair; electrocoagulation; postoperative pain; thermal injury; neuralgia
MeSH Terms: conditions — Hernia, Inguinal; Hyperthermia; Pain, Postoperative; Neuralgia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Electrocoagulation: Patients will undergo a standard procedure for inguinal hernia repair, with the use of electrocoagulation.
  Interventions: Procedure: Inguinal hernia repair
- No electrocoagulation: Patients will undergo a standard procedure for inguinal hernia repair, without the use of electrocoagulation.
  Interventions: Procedure: Inguinal hernia repair

INTERVENTIONS:
Procedure: Inguinal hernia repair — Standard procedure for inguinal hernia repair

SUMMARY:
Laparoscopic TAPP (transabdominal preperitoneal) hernia repair presents a minimally invasive surgical procedure, which tends to be a gold standard in a wide range of inguinal hernia operations. Postoperative neuralgia is a troublesome complication following TAPP, which occurs in 0.2-7% of patients. The most common cause of nerve injury is an inappropriate use of electrocoagulation or dangerous tissue dissection during TAPP. However, the association between electrocoagulation employment during TAPP and postoperative neuralgia has not been investigated properly until now.

The aim of the project is to compare postoperative pain (postoperative neuralgia) in patients undergoing TAPP inguinal hernia repair with/without the use of electrocoagulation.

DETAILED DESCRIPTION:
Worldwide, more than 20 million patients undergo inguinal hernia repair annually. Laparoscopic hernia repair presents a minimally invasive surgical procedure, which tends to be a gold standard for inguinal hernia repair. In comparison with open techniques of hernia repair, TAPP approach requires a totally different anatomic point of view. The operating surgeon must understand the basic principles and technical key points of TAPP in order to ensure satisfactory surgical outcomes and to prevent the occurrence of complications.

Postoperative neuralgia presents a troublesome complication following TAPP, which occurs in 0.2-7% of patients. Neuralgia is caused by intraoperative injury of genitofemoral, ilioinguinal, iliohypogastric or cutaneous femoris lateralis nerves (genitofemoral nerve being is the most often damaged). During TAPP, the most frequent causes of neural injury include clip application, inappropriate use of electrocoagulation or dangerous tissue dissection. At present, the employment of modern self-gripping meshes and tissue glues leave the use of electrocoagulation the main risk factor for potential nerve injury.

The aim of the proposed project is to evaluate postoperative pain (postoperative neuralgia) in patients undergoing TAPP inguinal hernia repair with/without the use of electrocoagulation. The assessment of the pain in the groin region will be performed on the 2nd and 7th postoperative day by means of clinical examination and by fulfilling the visual scale of pain. In patients showing clinical signs of postoperative neuralgia on the 7th postoperative day, clinical examination by an experienced neurologist will be performed.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* unilateral inguinal hernia
* no previous intraabdominal operations
* no history of neurological diseases

Exclusion Criteria:

* recurrent inguinal hernia
* bilateral inguinal hernia
* history of chronic pain syndrome
* preoperative ASA classification IV-V

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients indicated for an inguinal hernia surgical repair.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Postoperative neuralgia | 12 months
  The patients will assess the postoperative neuralgia in the groin area using a questionnaire with a 5-point scale (1-5). The value of 1 indicates no pain, value 5 indicates the highest possible imaginable pain, as assessed by the patients.

SECONDARY OUTCOMES:
Surgery time | 12 months
  The surgery time (skin to skin) will be measured in all patients (in minutes).
Scrotal hematoma | 12 months
  The presence of scrotal hematoma (yes/no) will be assessed in all patients.
Seroma | 12 months
  The presence of seroma (yes/no) will be assessed in all patients.

CONTACTS AND LOCATIONS:
Overall Officials: Petr Ostruszka, MD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava-Poruba, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: Undecided
The investigators have not decided to share the IPD with other researchers.

REFERENCES:
- [Background] Archvadze VSh, Chkhivadze TF, Giorgadze KI, Chanukvadze IM, Dzhikiia DT, Koberidze GI, Tsamalaidze AM. [Electrocoagulation in the surgery of inguinal hernias]. Khirurgiia (Mosk). 2006;(1):53-4. Russian. PMID 16482060
- [Background] Bittner R, Leibl B, Kraft K. [Laparoscopic hernia repair: prevention and therapy of complications]. Langenbecks Arch Chir Suppl Kongressbd. 1997;114:935-8. German. PMID 9574303
- [Background] Zohar Y, Sadov R, Strauss M, Djialdetti M. Ultrastructural study of peripheral nerve injury induced by monopolar and bipolar diathermy. Ann Otol Rhinol Laryngol. 1996 Sep;105(9):673-7. doi: 10.1177/000348949610500901. PMID 8800051
- [Background] Lee CH, Dellon AL. Surgical management of groin pain of neural origin. J Am Coll Surg. 2000 Aug;191(2):137-42. doi: 10.1016/s1072-7515(00)00319-7. PMID 10945356
- [Background] Bansal VK, Misra MC, Babu D, Victor J, Kumar S, Sagar R, Rajeshwari S, Krishna A, Rewari V. A prospective, randomized comparison of long-term outcomes: chronic groin pain and quality of life following totally extraperitoneal (TEP) and transabdominal preperitoneal (TAPP) laparoscopic inguinal hernia repair. Surg Endosc. 2013 Jul;27(7):2373-82. doi: 10.1007/s00464-013-2797-7. Epub 2013 Feb 7. PMID 23389072
- [Background] Singh AN, Bansal VK, Misra MC, Kumar S, Rajeshwari S, Kumar A, Sagar R, Kumar A. Testicular functions, chronic groin pain, and quality of life after laparoscopic and open mesh repair of inguinal hernia: a prospective randomized controlled trial. Surg Endosc. 2012 May;26(5):1304-17. doi: 10.1007/s00464-011-2029-y. Epub 2011 Nov 15. PMID 22083332
- [Background] Cesmebasi A, Yadav A, Gielecki J, Tubbs RS, Loukas M. Genitofemoral neuralgia: a review. Clin Anat. 2015 Jan;28(1):128-35. doi: 10.1002/ca.22481. Epub 2014 Nov 5. PMID 25377757